CLINICAL TRIAL: NCT04854369
Title: 68Ga-PSMA-11 Patients With Newly Diagnosed and Recurrent Prostate Cancer
Brief Title: 68Ga-PSMA-11 Patients With Newly Diagnosed and Recurrent Prostate Cancer (Firefly)
Acronym: Firefly
Status: No longer available | Type: Expanded Access
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-583
Record Dates: First submitted 2021-04-16; First posted 2021-04-22 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Prostatic Neoplasms; Prostatic Neoplasms, Castration-Resistant
Keywords: 68 Ga-PSMA-11; Prostate cancer; Metastatic prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Neoplasms, Castration-Resistant

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Drug: 68 Ga-PSMA-11 prepared using a PSMA-11 Sterile Cold Kit — The PSMA-11 Sterile Cold Kit is supplied as a kit for preparation of radiolabeled Gallium-68 PSMA-11 Injection, with 3 configurations (A, B or D) to accommodate the specificities of the 68Ge/68Ga generator that is used.

SUMMARY:
This is a prospective, Phase 2, single-center, open-label study of 68Ga-PSMA-11 PET scans in patients with biochemically recurrent prostate cancer or those diagnosed and untreated with high risk or very high risk localized prostate cancer, or oligometastatic (defined as three or fewer metastatic lesions on conventional imaging) prostate cancer (using NCCN classification for localized disease).

Approximately 300 patients are planned for enrollment in this study, divided into two cohorts. Cohort A will be 225 patients in the recurrent setting. Cohort B will be 75 patients in the up-front newly diagnosed setting.

After a screening period (6-week window), eligible patients will undergo baseline assessments as per the Schedule of Study Activities. Patients will receive a single dose of 68Ga-PSMA-11 and undergo a PET/CT or PET/MRI imaging study.

ELIGIBILITY:
Inclusion Criteria:

* Males greater than 18 years of age.
* Histologically proven adenocarcinoma of the prostate. Diagnosis must be stated in a pathology report and confirmed by the investigator.
* Patients must meet the criteria of one of the following cohorts:

Cohort A: (n=225) Biochemical recurrence; defined as any of the following:

* PSA ≥ 0.2 ng/mL and rising in at least two consecutive tests (at least one week apart) within 6 months of date of consent for patients treated with radical prostatectomy.
* PSA >2.0 ng/mL above the nadir and rising post-radiation (external beam or brachytherapy) +/- hormones, in at least 2 consecutive tests (at least one week apart) within 6 months of consent
* In patients with no prior definitive surgery or radiation, PSA ≥ 2 ng/mL greater than the post therapy nadir after androgen deprivation therapy.

Note: Patients whom have had more than one prior therapy, should be defined recurrent by their most recent therapy type. For patients who have had any ADT, are mCRPC, shall fall into that category for allocation and eligibility.

Cohort B: (n=75) No prior treatment defined as one of the following:

o Patient has primary diagnosis of "high risk" or "very high risk" localized prostate cancer, or regional prostate cancer (TxN1M0) or oligometastatic cancer (TxNXM1) with less than three metastatic lesions by conventional imaging) and has not received prior treatment.

Note: high risk/very high risk is denoted by Gleason 8-10, or PSA >20, or clinical stage T3a/T4 disease (see NCCN guidelines v1.2020).

Patients in this cohort must be considered candidates for initial definitive therapy at the time of study enrollment.

* Life expectancy of >6 months
* Patients should have a Comprehensive Metabolic Panel, PSA, and Testosterone drawn within 4 weeks of imaging

Exclusion Criteria:

* Claustrophobia or any other condition that would preclude PET/CT imaging.
* Patients with known metastatic prostate cancer, with 4 or more lesions on conventional imaging

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Alton O Sartor, MD, Principal Investigator — Tulane University
Locations (1):
- Tulane Medical Center, New Orleans, Louisiana, United States

REFERENCES:
- [Background] Cooperberg MR, Vickers AJ, Broering JM, Carroll PR. Comparative risk-adjusted mortality outcomes after primary surgery, radiotherapy, or androgen-deprivation therapy for localized prostate cancer. Cancer. 2010 Nov 15;116(22):5226-34. doi: 10.1002/cncr.25456. PMID 20690197
- [Background] Wallis CJD, Saskin R, Choo R, Herschorn S, Kodama RT, Satkunasivam R, Shah PS, Danjoux C, Nam RK. Surgery Versus Radiotherapy for Clinically-localized Prostate Cancer: A Systematic Review and Meta-analysis. Eur Urol. 2016 Jul;70(1):21-30. doi: 10.1016/j.eururo.2015.11.010. Epub 2015 Dec 15. PMID 26700655
- [Background] Lau WK, Bergstralh EJ, Blute ML, Slezak JM, Zincke H. Radical prostatectomy for pathological Gleason 8 or greater prostate cancer: influence of concomitant pathological variables. J Urol. 2002 Jan;167(1):117-22. PMID 11743287
- [Background] Thompson IM, Valicenti RK, Albertsen P, Davis BJ, Goldenberg SL, Hahn C, Klein E, Michalski J, Roach M, Sartor O, Wolf JS Jr, Faraday MM. Adjuvant and salvage radiotherapy after prostatectomy: AUA/ASTRO Guideline. J Urol. 2013 Aug;190(2):441-9. doi: 10.1016/j.juro.2013.05.032. Epub 2013 May 21. PMID 23707439
- [Background] Moreira DM, Presti JC Jr, Aronson WJ, Terris MK, Kane CJ, Amling CL, Freedland SJ. Natural history of persistently elevated prostate specific antigen after radical prostatectomy: results from the SEARCH database. J Urol. 2009 Nov;182(5):2250-5. doi: 10.1016/j.juro.2009.07.022. Epub 2009 Sep 16. PMID 19758614
- [Background] Stephenson AJ, Scardino PT, Kattan MW, Pisansky TM, Slawin KM, Klein EA, Anscher MS, Michalski JM, Sandler HM, Lin DW, Forman JD, Zelefsky MJ, Kestin LL, Roehrborn CG, Catton CN, DeWeese TL, Liauw SL, Valicenti RK, Kuban DA, Pollack A. Predicting the outcome of salvage radiation therapy for recurrent prostate cancer after radical prostatectomy. J Clin Oncol. 2007 May 20;25(15):2035-41. doi: 10.1200/JCO.2006.08.9607. PMID 17513807
- [Background] Ajib K, Zanaty M, Alnazari M, Rajih E, Hueber PA, Mansour M, Valdivieso R, Negrean C, Karakiewicz PI, Taussky D, Delouya G, El-Hakim A, Zorn KC. Functional and oncological outcomes of salvage external beam radiotherapy following robot-assisted radical prostatectomy in a Canadian cohort. Can Urol Assoc J. 2018 Feb;12(2):45-49. doi: 10.5489/cuaj.4641. Epub 2017 Dec 1. PMID 29381466
- [Background] Freedland SJ, Rumble RB, Finelli A, Chen RC, Slovin S, Stein MN, Mendelson DS, Wackett C, Sandler HM; American Society of Clinical Oncology. Adjuvant and salvage radiotherapy after prostatectomy: American Society of Clinical Oncology clinical practice guideline endorsement. J Clin Oncol. 2014 Dec 1;32(34):3892-8. doi: 10.1200/JCO.2014.58.8525. Epub 2014 Nov 3. PMID 25366677
- [Background] Fendler WP, Calais J, Eiber M, Flavell RR, Mishoe A, Feng FY, Nguyen HG, Reiter RE, Rettig MB, Okamoto S, Emmett L, Zacho HD, Ilhan H, Wetter A, Rischpler C, Schoder H, Burger IA, Gartmann J, Smith R, Small EJ, Slavik R, Carroll PR, Herrmann K, Czernin J, Hope TA. Assessment of 68Ga-PSMA-11 PET Accuracy in Localizing Recurrent Prostate Cancer: A Prospective Single-Arm Clinical Trial. JAMA Oncol. 2019 Jun 1;5(6):856-863. doi: 10.1001/jamaoncol.2019.0096. PMID 30920593
- [Background] Calais J, Ceci F, Eiber M, Hope TA, Hofman MS, Rischpler C, Bach-Gansmo T, Nanni C, Savir-Baruch B, Elashoff D, Grogan T, Dahlbom M, Slavik R, Gartmann J, Nguyen K, Lok V, Jadvar H, Kishan AU, Rettig MB, Reiter RE, Fendler WP, Czernin J. 18F-fluciclovine PET-CT and 68Ga-PSMA-11 PET-CT in patients with early biochemical recurrence after prostatectomy: a prospective, single-centre, single-arm, comparative imaging trial. Lancet Oncol. 2019 Sep;20(9):1286-1294. doi: 10.1016/S1470-2045(19)30415-2. Epub 2019 Jul 30. PMID 31375469
- [Background] Perera M, Papa N, Christidis D, Wetherell D, Hofman MS, Murphy DG, Bolton D, Lawrentschuk N. Sensitivity, Specificity, and Predictors of Positive 68Ga-Prostate-specific Membrane Antigen Positron Emission Tomography in Advanced Prostate Cancer: A Systematic Review and Meta-analysis. Eur Urol. 2016 Dec;70(6):926-937. doi: 10.1016/j.eururo.2016.06.021. Epub 2016 Jun 28. PMID 27363387
- [Background] Fendler WP, Eiber M, Beheshti M, Bomanji J, Ceci F, Cho S, Giesel F, Haberkorn U, Hope TA, Kopka K, Krause BJ, Mottaghy FM, Schoder H, Sunderland J, Wan S, Wester HJ, Fanti S, Herrmann K. 68Ga-PSMA PET/CT: Joint EANM and SNMMI procedure guideline for prostate cancer imaging: version 1.0. Eur J Nucl Med Mol Imaging. 2017 Jun;44(6):1014-1024. doi: 10.1007/s00259-017-3670-z. PMID 28283702
- [Background] Hope TA, Goodman JZ, Allen IE, Calais J, Fendler WP, Carroll PR. Metaanalysis of 68Ga-PSMA-11 PET Accuracy for the Detection of Prostate Cancer Validated by Histopathology. J Nucl Med. 2019 Jun;60(6):786-793. doi: 10.2967/jnumed.118.219501. Epub 2018 Dec 7. PMID 30530831
- [Background] Afshar-Oromieh A, Malcher A, Eder M, Eisenhut M, Linhart HG, Hadaschik BA, Holland-Letz T, Giesel FL, Kratochwil C, Haufe S, Haberkorn U, Zechmann CM. PET imaging with a [68Ga]gallium-labelled PSMA ligand for the diagnosis of prostate cancer: biodistribution in humans and first evaluation of tumour lesions. Eur J Nucl Med Mol Imaging. 2013 Apr;40(4):486-95. doi: 10.1007/s00259-012-2298-2. Epub 2012 Nov 24. PMID 23179945